CLINICAL TRIAL: NCT01879449
Title: Prevalence of Spasticity in Veterans Living in a Long-term Care Facility
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Allergan (Industry); Merz North America, Inc. (Industry)
Responsible Party: Principal Investigator, David Charles, Professor and Vice-Chair, Department of Neurology, Vanderbilt University
Other Study IDs: 110470VU; VUMC38674-R (Other Grant/Funding Number: Merz Pharma); VUMC35131-R (Other Grant/Funding Number: Allergan, Inc.)
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Spasticity
Keywords: Spasticity; Veterans; Prevalence
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to conduct a feasibility survey of the prevalence of spasticity at a single long-term care facility for veterans and their spouses in Murfreesboro, Tennessee. These data will be used to strengthen a future grant application to the Department of Defense in response to their ongoing Traumatic Brain Injury initiative.

DETAILED DESCRIPTION:
The goal of this feasibility survey is to determine the prevalence of spasticity that interferes with care or function at the Tennessee State Veterans Home (TSVH), which is a long-term care facility for veterans and their spouses in Murfreesboro, Tennessee. In order to accomplish this goal, each of the 140 residents will be examined by the principal investigator and a medical record review will be performed; also, each patient and their medical decision-maker (if applicable), direct caregiver, and treating physician will be surveyed in order to further elucidate the barriers to treatment in this population. All consenting residents of the TSVH will be examined, but the data will be separated prior to analysis based on whether the resident is a veteran or a veteran's relative.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects of any race, aged 18 and above.
* Reside at the Tennessee State Veterans Home

Exclusion Criteria:

* Subjects for whom it is felt that participation in the study would cause medical harm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nursing home residents
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Spasticity diagnosis | Up to three months after consent is obtained
  There is no biomarker for spasticity. Therefore, the diagnosis will be made on physician impression. A neurologist trained in movement disorders will examine each consented patient to determine if they have spasticity. The severity of the veteran's spasticity will be documented, including the following measures: presence of fixed contractures and presence of pain on movement.

SECONDARY OUTCOMES:
Spasticity treatment awareness and preferences survey | Up to three months after consent is obtained
  The investigators will use a structured interview to assess each subject's level of awareness of available treatments for spasticity. Subjects will be asked if they are aware of specific treatments for spasticity and asked to answer "yes" or "no".
  This interview is also designed to capture subjects' spasticity treatment preferences. Subjects will be asked if they are interested in receiving a variety of available spasticity treatments and asked to answer "yes," "no," or "maybe".

CONTACTS AND LOCATIONS:
Overall Officials: David Charles, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Tennessee State Veterans Home, Murfreesboro, Tennessee, United States